CLINICAL TRIAL: NCT01885403
Title: Non-Invasive Pulmonary Monitoring in Patients With Cardiogenic Pulmonary Congestion and Edema
Brief Title: Acute Congestive Heart Failure
Acronym: AcuteCHF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Collaborators: Philips Technology Aachen Germany (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CTC-A 12-117
Record Dates: First submitted 2013-06-20; First posted 2013-06-25 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Acute Decompensated Heart Failure (ADHF); Acute Cardiogenic Pulmonary Edema (ACPE)
Keywords: Acute Cardiogenic Pulmonary Edema,; Acute Decompensated Heart Failure,; BiLevel Positive Airway Pressure,; Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Respiratory Parameters Measurements (Experimental)
  Interventions: Device: non-invasive respiratory parameter measurements

INTERVENTIONS:
Device: non-invasive respiratory parameter measurements
  Other Names: Philips Respironics BiPAP Synchrony, Bioimpedance ImpediMed- SFB7

SUMMARY:
The aim of the study is to determine the feasibility of collecting respiratory parameters during recompensation following ADHF (Acute Decompensated Heart Failure)with non-invasive measurements. This could lead to a better understanding of how respiratory parameters may change during re-compensation therapy and could also be a comfortable method for patients.

DETAILED DESCRIPTION:
The study is designed as a single-center, open, interventional, observational study according to clause §23b of the German Medical Device Act (MPG). The study will recruit 50 patients suffering from cardiogenic pulmonary congestion and edema including ambulant patients and patients of intensive care.

We will investigate whether respiratory parameters during re-compensation are related to the therapy effects and changes in pulmonary congestion status. This study will collect data in an observational and clinical setting in the re-compensation phase of ADHF.

Correlation between measured lung and respiratory parameters and standard clinical parameters characterizing stages of re-compensation will be undertaken. Standard clinical parameters may include diuretics and other cardiac medication dose frequency, weight, heart rate, respiratory rate, chest x-rays (when routinely performed), symptoms such as shortness of breath or fatigue, biomarkers such as brain natriuretic peptide (BNP), stroke volume, cardiac output, and oxygen requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, ages 18-75
2. Able and willing to provide written informed consent or not able to give informed consent because of mechanical respiration
3. Diagnosis of acute or chronic decompensated heart failure with pulmonary congestion or edema
4. Systolic blood pressure >80 mm Hg at time of enrollment
5. Resting pulse oximetry (SpO2) at the time of enrollment of at least 88% at 21% iron oxides (FeO2)
6. Agreement to be measured with the study devices according to study protocol by patient or legal representative
7. Left ventricular ejection fraction (LVEF) < 40% in 3D- Echocardiography

Exclusion Criteria:

1. Active participation in another interventional research study
2. Surgery of the upper airway, nose, sinus or middle ear within the last 90 days
3. Major medical or psychiatric condition that would interfere with the demands of the study or the ability to complete the study. For example, severe unstable chronic lung disease such as obstructive (FEV1/FVC ≤ 30%), or restrictive (FVC < 50% predicted) lung disease, neuromuscular disease, cancer, or renal failure
4. Unable to use PAP therapies due to physical issues (e.g. facial structural abnormalities) or cognitive issues (e.g. dementia)
5. Participants in whom positive airway pressure (PAP) therapy is medically contraindicated.
6. Uncontrolled hypertension (systolic ≥200 mm Hg/diastolic ≥120 mm Hg)
7. Pregnancy
8. Lactation
9. Implanted pacemaker / Cardiac Resynchronization Therapy (CRT) / implantable cardioverter-defibrillator (ICD) except for Medtronic devices with Opti Vol Algorithm
10. Incompetent patients or patients who, in the judgment of the investigator, are too unstable or are otherwise not capable of performing study procedures
11. Post-partum cardiomyopathy
12. Hypertrophic
13. Primary mitral valve stenosis
14. Patients requiring more than 50% supplemental oxygen or patients requiring more than 4 lpm oxygen
15. Patients with persistent ventricular arrhythmias (Premature ventricular coupling, periods of ventricular tachycardia)
16. Patients chronically classified (prior to admission) as New York Heart Association (NYHA) Class IV or American Heart Association Class D heart failure
17. Patients with glomerular filtration rate (GFR) <30 or obligatory dialysis
18. Resting respiratory rate >30 breaths per minute
19. Patients requiring mechanical ventilation or patients with an artificial airway (endotracheal or tracheostomy tube)
20. Patients with carbon monoxide toxicity
21. Patients with severe sepsis (defined as also an organ dysfunction due to an infection according to the Guidelines of the German Association of Sepsis, February 2010)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Correlation between current standard clinical assessment of re-compensation and measured respiratory parameters | about 3 months
  stationary as well as ambulant patients with acute decompensation receive clinical standard measurements and will be measured with the help of non- invasive technology such as respiratory profile and gaz analysis, bioimpedance spectroscopy. Patients will be measured at baseline and 2 times at ward if applicable and at 3 months follow up visit. Measurements will take 1:30 hours per visit.

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Schröder, MD, Principal Investigator — Department of Cardiology, Pneumology, Angiology and Intensive Care, Internal Medicine I (MK I), University Hospital Aachen (UKA)
Locations (1):
- University Hospital of Aachen, Department of Cardiology, Aachen, Northrhine-Westfalia, Germany